CLINICAL TRIAL: NCT03180619
Title: A Phase 2, Open-label Study to Evaluate the Safety and Efficacy of Switching to Tenofovir Alafenamide (TAF) From Tenofovir Disoproxil Fumarate (TDF) and/or Other Oral Antiviral Treatment (OAV) in Virologically Suppressed Chronic Hepatitis B Subjects With Renal and/or Hepatic Impairment
Brief Title: Study to Evaluate the Safety and Efficacy of Switching to Tenofovir Alafenamide (TAF) From Tenofovir Disoproxil Fumarate (TDF) and/or Other Oral Antiviral Treatment (OAV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-320-4035; 2016-004625-16 (EudraCT Number)
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Results first posted 2020-04-09 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Renal Impairment): Moderate or Severe Renal Impairment (Experimental): Participants with chronic hepatitis B (CHB) and moderate or severe renal impairment who were virologically suppressed and taking tenofovir disoproxil fumarate (TDF), a TDF-containing anti-hepatitis B virus (HBV) regimen, or other oral antivirals (OAVs), will switch to tenofovir alafenamide (TAF) and receive TAF 25 milligram (mg) tablet once daily orally for 96 weeks.
  Interventions: Drug: TAF
- Part A (Renal Impairment): End Stage Renal Disease (Experimental): Participants with CHB and end stage renal disease who were virologically suppressed and taking TDF, a TDF-containing anti-HBV regimen, or OAVs, will switch to TAF and receive TAF 25 mg tablet once daily orally for 96 weeks.
  Interventions: Drug: TAF
- Part B: Hepatic Impairment (Experimental): Participants with CHB and moderate or severe hepatic impairment who were virologically suppressed and taking TDF, a TDF-containing anti-HBV regimen, or OAVs, will switch to TAF and receive TAF 25 mg tablet once daily orally for 96 weeks.
  Interventions: Drug: TAF

INTERVENTIONS:
Drug: TAF — Tablet administered orally once daily
  Other Names: Vemlidy®

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability and virologic response of tenofovir alafenamide (TAF) in virologically suppressed chronic hepatitis B participants with renal and/or hepatic impairment.

ELIGIBILITY:
Key Inclusion Criteria:

All Participants (Parts A and B):

* Adult male or non-pregnant female individuals
* Documented evidence of chronic HBV infection
* Alanine aminotransferase (ALT) ≤ 10 × upper limit of normal (ULN)

Part A Only (renal impairment):

* Maintained on TDF and/or other OAV treatment(s) for CHB for at least 48 weeks and with viral suppression (HBV deoxyribonucleic acid [DNA] < lower limit of quantitation [LLOQ]) for ≥ 6 months prior to screening

  * All individuals must have HBV DNA < 20 International units per milliliter (IU/mL) at screening by central laboratory
  * Both Hepatitis B e-Antigen (HBeAg) positive and negative individuals are eligible to participate
* Moderate renal impairment (30 milliliters per minute [mL/min] ≤ estimated glomerular filtration rate by the cockcroft-gault formula [eGFRcg] ≤ 59 mL/min), severe renal impairment (15 mL/min ≤ eGFRcg < 30 mL/min) or end stage renal disease (ESRD) (eGFR < 15 mL/min) maintained on hemodialysis (HD)
* Stable renal function (for participants with moderate or severe impairment): serum creatinine measured at least once within three months prior to screening. The measurement difference between the value measured within three months prior to screening versus the screening value must be ≤ 25% of the screening value

Part B Only (hepatic impairment):

* Maintained on TDF and/or other OAV(s) for CHB for at least 48 weeks and with viral suppression (HBV DNA < LLOQ) for ≥ 6 months prior to screening

  * All individuals must have HBV DNA < 20 IU/mL at screening by central laboratory
  * Both HBeAg positive and negative individuals are eligible to participate
* Child-pugh-turcotte (CPT) score of 7-12 (inclusive) OR a past history of CPT score ≥ 7 and any CPT score ≤ 12 at screening
* eGFRCG ≥ 30 mL/min using the Cockcroft-Gault equation

Key Exclusion Criteria:

All Individuals (Parts A & B):

* Women who are breastfeeding or who believe they may wish to become pregnant during the course of the study
* Males and females of reproductive potential who are unwilling to use an "effective", protocol-specified method(s) of contraception during the study
* Co-infection with hepatitis C virus (HCV), human immunodeficiency virus (HIV), or hepatitis D virus (HDV)
* Prior Interferon (IFN) use within 6 months of screening
* Evidence of hepatocellular carcinoma
* Received solid organ or bone marrow transplant
* Significant cardiovascular, pulmonary, or neurological disease
* Malignancy within 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc.). Individuals under evaluation for possible malignancy are not eligible
* Currently receiving therapy with immunomodulators (e.g. corticosteroids), nephrotoxic agents, or agents capable of modifying renal excretion
* Known hypersensitivity to study drugs, metabolites, or formulation excipients
* Current alcohol or substance abuse judged by the investigator to potentially interfere with individual's compliance
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the individual unsuitable for the study or unable to comply with dosing requirements.

Part A Only (Renal Impairment):

* Current or historical evidence of clinical hepatic decompensation (e.g., ascites, encephalopathy or variceal hemorrhage)
* Abnormal hematological and biochemical parameters, including:

  * Hemoglobin < 9 grams per deciliter (g/dL)
  * Absolute neutrophil count < 750/cubic millimeter (mm^3)
  * Platelets ≤ 50,000/mm^3
  * Aspartate aminotransferase (AST) > 10 × ULN
  * Albumin < 3.0 g/dL
  * Total bilirubin > 2.5 × ULN
  * International normalized ratio of prothrombin time (INR) > 1.5 × ULN (unless stable on anticoagulant regimen)
* Individuals with ESRD (i.e. eGFRcg < 15 mL/min) not on HD, or those on other forms of renal replacement therapy (i.e. peritoneal dialysis)

Part B Only (Hepatic Impairment):

* Active variceal bleeding within 6 months or prior placement of a portosystemic shunt (such as transjugular intrahepatic portosystemic shunt [TIPS])
* History of hepatorenal syndrome, hepatopulmonary syndrome, Grade 3 or Grade 4 hepatic encephalopathy, or spontaneous bacterial peritonitis within 6 months of screening
* Grade 2 hepatic encephalopathy at screening
* Model for end-stage liver disease (MELD) score ≥ 30
* Abnormal hematological and biochemical parameters, including

  * Absolute neutrophil count < 750/mm^3
  * Platelets < 30,000/mm^3
  * Hemoglobin < 8.0 g/dL

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2020-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (30):
- United States (4):
  - Coalition of Inclusive Medicine, Los Angeles, California
  - Silicon Valley Research Institute, Inc, San Jose, California
  - Henry Ford Health System, Detroit, Michigan
  - Harborview Medical Center, Seattle, Washington
- Canada (5):
  - University of Calgary Liver Unit, Calgary
  - Centre de Recherche du Centre Hospitalier de l'Universite de Montreal, Montreal
  - University Health Network,Toronto general Hospital,Toronto centre for liver disease, Toronto
  - Toronto Liver Centre, Toronto
  - (G.I.R.I.) GI Research Institute, Vancouver
- Hong Kong (3):
  - Prince of Wales Hospital, Shatin, NT
  - Princess Margaret Hospital, Kowloon
  - Alice Ho Miu Ling Nethersole Hospital, Tai Po
- Italy (3):
  - U.O. Medicina Generale Epatologia IRCCS Humanitas Centro di Ricerca Traslazionale in Epatologia, Rozzano, Milan
  - Dipartimento di Scienze Mediche e Chirurgiche (DIMEC) AOU Policlinico S.Orsola-Malpighi di Bologna, Bologna
  - UOC Gastroenterol-Epatol.-Fondazione IRCCS Ca Granda, Milan
- Auckland Clinical Studies, Grafton, Auckland, New Zealand
- South Korea (4):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Asan Medical Center, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
- Taiwan (8):
  - Changhua Christian Hospital, Changhua
  - Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans Genl Hosp, Taichung
  - National Taiwan University Hospital, Taipei
  - Veterans General Hospital-Taipei, Taipei
  - Chang Gung Medical Foundation, Linkou Chang Gung Memorial Hospital, Taoyuan
- United Kingdom (2):
  - Nottingham University Hospital, London
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Lim YS, Lin CY, Heo J, Bae H, Chuang WL, Hui AJ, et al. Safety and Efficacy of Switching to Tenofovir Alafenamide in Virally Suppressed Chronic Hepatitis B Patients With Hepatic Impairment: Week-48 Results From a Phase 2 Open-label Study [Poster SAT442]. The Digital International Liver Congress (ILC); 2020 27-29 August.
- [Result] Janssen HLA, Lampertico P, Chen CY, Heo J, Fournier C, Ahn SH, et al. Safety and Efficacy of Switching to Tenofovir Alafenamide in Virally Suppressed Chronic Hepatitis B Patients With Renal Impairment: Week-48 Results From a Phase 2 Open-label Study [Poster SAT429]. The Digital International Liver Congress (ILC); 2020 27-29 August.
- [Result] Lim YS, Lampertico P, Bae H, Chuang WL, Heo J, Huang YH, et al. Switching From Tenofovir Disoproxil Fumarate or Other Oral Antiviral Therapy to Tenofovir Alafenamide in Virally Suppressed Chronic Hepatitis B Patients With Hepatic Impairment: Week 24 Efficacy and Safety Results From a Phase 2 Open-label Study [Poster 501]. AASLD: The Liver Meeting; 2019 08-12 November; Boston, MA.
- [Result] Janssen HLA, Lim YS, Gane EJ, Fournier C, Ahn SH, Tsang O, et al. Efficacy and Safety of Switching to Tenofovir Alafenamide in Virally Suppressed Chronic Hepatitis B Patients With Renal Impairment: Week 24 Results From a Phase 2 Open-label Study [Poster 483]. AASLD: The Liver Meeting; 2019 08-12 November; Boston, MA.
- [Derived] Liu CJ, Lim YS, Chen CY, Chen CH, Huang YH, Lin CY, Lin CC, Yu ML, Abramov F, Yee LJ, Duan R, Flaherty JF, Su WW, Yang SS, Janssen HLA, Chuang WL. Switching to tenofovir alafenamide in virally-suppressed chronic hepatitis B patients with renal/hepatic impairment: Phase 2 study sub-analysis from Taiwan. J Formos Med Assoc. 2025 Jul 30:S0929-6646(25)00390-0. doi: 10.1016/j.jfma.2025.07.023. Online ahead of print. PMID 40744841
- [Derived] Janssen HLA, Lim YS, Lampertico P, Heo J, Chen CY, Fournier C, Tsang TYO, Bae H, Chen CH, Coffin CS, Ahn SH, Trinh H, Flaherty JF, Abramov F, Zhao Y, Liu Y, Lau A, German P, Chuang WL, Agarwal K, Gane E. Switching to tenofovir alafenamide in patients with virologically suppressed chronic hepatitis B and renal or hepatic impairment: final week 96 results from an open-label, multicentre, phase 2 study. Lancet Gastroenterol Hepatol. 2024 Aug;9(8):718-733. doi: 10.1016/S2468-1253(24)00096-7. Epub 2024 Jun 17. PMID 38901444

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Asia Pacific, North America, New Zealand and Europe. The first participant was screened on 29 June 2017. The last study visit occurred on 04 September 2020.
Pre-assignment Details: 147 participants were screened.
Groups:
- Part A (Renal Impairment): Moderate or Severe Renal Impairment: Participants with chronic hepatitis B (CHB) and moderate or severe renal impairment who were virologically suppressed and took tenofovir disoproxil fumarate (TDF), a TDF-containing anti-hepatitis B virus (HBV) regimen, or other oral antivirals (OAVs), switched to tenofovir alafenamide (TAF) and received TAF 25 mg tablet once daily orally for 96 weeks.
- Part A (Renal Impairment): End Stage Renal Disease: Participants with CHB and end stage renal disease who were virologically suppressed and took TDF, a TDF-containing anti-HBV regimen, or OAVs, switched to TAF and received TAF 25 mg tablet once daily orally for 96 weeks.
- Part B: Hepatic Impairment: Participants with CHB and moderate or severe hepatic impairment who were virologically suppressed and took TDF, a TDF-containing anti-HBV regimen, or OAVs, switched to TAF and received TAF 25 mg tablet once daily orally for 96 weeks.
Period: Overall Study
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Started | 78 | 15 | 31
Completed | 67 | 14 | 25
Not Completed | 11 | 1 | 6
Not completed — Withdrew Consent | 5 | 0 | 2
Not completed — Death | 2 | 1 | 2
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Investigator's discretion | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Part A (Renal Impairment): Moderate or Severe Renal Impairment: Participants with CHB and moderate or severe renal impairment who were virologically suppressed and taking TDF, a TDF-containing anti-HBV regimen, or other OAVs, switched to TAF and received TAF 25 mg tablet once daily orally for 96 weeks.
- Part A (Renal Impairment): End Stage Renal Disease: Participants with CHB and end stage renal disease who were virologically suppressed and taking TDF, a TDF-containing anti-HBV regimen, or OAVs, switched to TAF and received TAF 25 mg tablet once daily orally for 96 weeks.
- Part B: Hepatic Impairment: Participants with CHB and moderate or severe hepatic impairment who were virologically suppressed and taking TDF, a TDF-containing anti-HBV regimen, or OAVs, switched to TAF and received TAF 25 mg tablet once daily orally for 96 weeks.
- Total: Total of all reporting groups
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment | Total
Number analyzed (Participants) | 78 | 15 | 31 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10.1) | 54 (12.8) | 55 (10.8) | 61 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 3 | 10 | 34
  Male | 57 | 12 | 21 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 1 | 1
  Ethnicity: Not Hispanic or Latino | 78 | 15 | 30 | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 59 | 13 | 25 | 97
  Race: Black or African American | 3 | 0 | 1 | 4
  Race: Native Hawaiian or Pacific Islander | 0 | 2 | 0 | 2
  Race: White | 15 | 0 | 4 | 19
  Race: Other | 1 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 0 | 2 | 0 | 2
  Canada | 22 | 0 | 3 | 25
  South Korea | 12 | 3 | 5 | 20
  Hong Kong | 14 | 1 | 2 | 17
  United States | 3 | 0 | 7 | 10
  Taiwan | 13 | 9 | 11 | 33
  Italy | 13 | 0 | 2 | 15
  United Kingdom | 1 | 0 | 1 | 2
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: Units/Liter (U/L)] | 20 (9.6) | 14 (5.2) | 28 (12.4) | 21 (10.8)
ALT Level Based on Central Lab Normal Range [Count of Participants; unit: Participants] — Central laboratory upper limit of normal (ULN) for ALT were as follows: ≤ 43 U/L for males aged 18 to < 69 years and ≤ 35 U/L for males aged ≥ 69 years; ≤ 34 U/L for females aged 18 to < 69 years and ≤ 32 U/L for females aged ≥ 69 years.
  Participants
    ≤ ULN | 75 | 15 | 27 | 117
    > ULN - 5xULN | 3 | 0 | 4 | 7
    > 5xULN | 0 | 0 | 0 | 0
ALT Level Based on 2018 American Association for the Study of Liver Diseases (AASLD) Normal Range [Count of Participants; unit: Participants] — The ULN for ALT using the 2018 AASLD normal range was 25 U/L for females and 35 U/L for males.
  Participants
    ≤ ULN | 73 | 15 | 21 | 109
    > ULN - 5xULN | 5 | 0 | 10 | 15
    > 5xULN | 0 | 0 | 0 | 0
Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Categories [Count of Participants; unit: Participants]
  < 20 IU/mL | 77 | 14 | 31 | 122
  ≥ 20 IU/mL - < 69 IU/mL | 0 | 1 | 0 | 1
  ≥ 69 IU/mL | 1 | 0 | 0 | 1
Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFRcg) [Mean (Standard Deviation); unit: milliliter/minute (mL/min)] — GFR is a measure of the rate at which blood is filtered by the kidney. Cockcroft-Gault is an equation (calculation) used to estimate GFR based on serum creatinine, weight, and gender. eGFRcg = (140 - age in years) * (body weight in kg) * (0.85 if female) divided by 72 * serum creatinine in mg/dL.
  milliliter/minute (mL/min) | 45.5 (10.89) | 7.8 (2.63) | 98.8 (33.94) | 54.3 (34.16)
Hip Bone Mineral Density (BMD) Status [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Hip Dual-Energy X-Ray Absorptiometry (DXA) Analysis Set included all participants who were enrolled and received at least 1 dose of study drug and had non-missing baseline hip BMD values.
  Participants
    number analyzed (Participants) | 77 | 15 | 31 | 123
    Normal (T-score ≥ -1.0) | 34 | 3 | 18 | 55
    Osteopenia (-2.5 ≤ T-score < -1.0) | 36 | 5 | 12 | 53
    Osteoporosis (T-score < -2.5) | 7 | 7 | 1 | 15
Spine BMD Status [Count of Participants; unit: Participants] — Measure Analysis Population Description: The Spine DXA Analysis Set included all participants who were enrolled and received at least 1 dose of study drug and had non-missing baseline spine BMD values.
  Participants
    Normal (T-score ≥ -1.0) | 37 | 5 | 16 | 58
    Osteopenia (-2.5 ≤ T-score < -1.0) | 22 | 7 | 9 | 38
    Osteoporosis (T-score < -2.5) | 19 | 3 | 6 | 28
Hepatitis s-Antigen (HBsAg) (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 2.51 (0.782) | 2.72 (1.405) | 1.90 (1.169) | 2.38 (1.012)
Hepatitis B e Antigen/Antibody (HBeAg/HBeAb) Status [Count of Participants; unit: Participants]
  Positive/Negative | 13 | 3 | 3 | 19
  Positive/Positive | 0 | 0 | 0 | 0
  Negative/Negative | 15 | 1 | 10 | 26
  Negative/Positive | 50 | 11 | 18 | 79
FibroTest® Score [Mean (Standard Deviation); unit: units on a scale] — The FibroTest® score is used to assess liver fibrosis. Scores range from 0.00 to 1.00, with higher scores indicating a greater degree of fibrosis Population: Participants in Safety Analysis Set with available data were analyzed.
  units on a scale
    number analyzed (Participants) | 77 | 15 | 31 | 123
    (all) | 0.53 (0.199) | 0.37 (0.199) | 0.75 (0.206) | 0.57 (0.231)
Child-Pugh-Turcotte (CPT) Score [Mean (Standard Deviation); unit: units on a scale] — CPT scores grade the severity of cirrhosis and are used to determine the need for liver transplantation. Scores can range from 5 to 15, with higher scores indicating a greater severity of disease. Population: Participants in the Full Analysis Set only from Part B (Hepatic Impairment) were analyzed.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 31 | 31
    (all) |  |  | 6 (1.7) | 6 (1.7)
Model for End-Stage Liver Disease (MELD) Score [Mean (Standard Deviation); unit: units on a scale] — MELD scores are used to assess prognosis and suitability for liver transplantation. Scores can range from 6 to 40, with higher scores indicating greater disease severity. Population: Participants in Full Analysis Set only from Part B (Hepatic Impairment) were analyzed.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 31 | 31
    (all) |  |  | 10.7 (3.40) | 10.7 (3.40)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Virologic Response (Plasma Hepatitis B Virus [HBV] Deoxyribonucleic Acid [DNA] < 20 IU/mL) at Week 24
Description: The percentage of participants with HBV DNA < 20 IU/mL at Week 24 was determined by the Missing = Failure (M = F) approach.
Time Frame: Week 24
Population: The Full Analysis Set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants | 97.4 | 100.0 | 100.0

2. Primary Outcome: Percentage of Participants Who Experienced Graded Treatment-Emergent Adverse Events (AEs) at Week 24
Description: Treatment-emergent AEs were defined as:
  * Any AEs with an onset date on or after the study drug start date and no later than the study drug stop date + 3 days after permanent discontinuation of study drug;
  * Any AEs with onset date on or after the study drug start date for those who have not permanently discontinued study drug;
  * Any AEs leading to premature discontinuation of study drug.
  The most severe graded AE from all tests was counted for each participant.
Time Frame: Week 24
Population: The Safety Analysis Set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants
  Any Treatment-emergent AEs | 53.8 | 73.3 | 54.8
  Grade 3 and Above Treatment-emergent AEs | 6.4 | 13.3 | 6.5

3. Primary Outcome: Percentage of Participants Who Experienced Graded Treatment-Emergent Laboratory Abnormalities at Week 24
Description: Graded treatment-emergent laboratory abnormalities were defined as values that increased at least 1 toxicity grade from baseline at any postbaseline visit, up to and including the date of last dose of study drug + 3 days for participants who permanently discontinued study drug or the last available date in the database snapshot for participants who were on treatment at the time of the analysis.
  The most severe graded abnormality from all tests was counted for each participant.
Time Frame: Week 24
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants
  Any Graded Laboratory Abnormality | 96.2 | 100.0 | 90.3
  Grade 3 and Above Laboratory Abnormality | 11.5 | 46.7 | 48.4

4. Secondary Outcome: Percentage of Participants Who Experienced Graded Treatment-Emergent AEs at Week 48
Description: Treatment-emergent AEs were defined as: Any AEs with an onset date on or after the study drug start date and no later than the study drug stop date + 3 days after permanent discontinuation of study drug; Any AEs with onset date on or after the study drug start date for those who have not permanently discontinued study drug; Any AEs leading to premature discontinuation of study drug. The most severe graded AE from all tests was counted for each participant.
Time Frame: Week 48
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants
  Any Treatment-emergent AE | 71.8 | 86.7 | 71.0
  Grade 3 and Above Treatment-emergent AEs | 15.4 | 20.0 | 12.9

5. Secondary Outcome: Percentage of Participants Who Experienced Graded Treatment-Emergent AEs at Week 96
Description: as for outcome 4
Time Frame: Week 96
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants
  Any Treatment-emergent AEs | 74.4 | 100.0 | 77.4
  Grade 3 and Above treatment-emergent AEs | 17.9 | 26.7 | 25.8

6. Secondary Outcome: Percentage of Participants Who Experienced Graded Treatment-Emergent Laboratory Abnormalities at Week 48
Description: as for outcome 3
Time Frame: Week 48
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants
  Any Graded Laboratory Abnormality | 96.2 | 100.0 | 90.3
  Grade 3 | 12.8 | 40.0 | 41.9
  Grade 4 | 0 | 26.7 | 9.7

7. Secondary Outcome: Percentage of Participants Who Experienced Graded Treatment-Emergent Laboratory Abnormalities at Week 96
Description: Graded treatment-emergent laboratory abnormalities were defined as values that increased at least 1 toxicity grade from baseline at any post-baseline visit, up to and including the date of last dose of study drug + 3 days for participants who permanently discontinued study drug or the last available date in the database snapshot for participants who were on treatment at the time of the analysis. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: Week 96
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of particpants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of particpants
  Any Graded Laboratory Abnormality | 96.2 | 100.0 | 100.0
  Grade 3 | 15.4 | 46.7 | 41.9
  Grade 4 | 1.3 | 26.7 | 12.9

8. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFRcg) in Participants With Moderate or Severe Renal Impairment and Hepatically Impaired Participants at Week 24
Description: GFR is a measure of the rate at which blood is filtered by the kidney. Cockcroft-Gault is an equation (calculation) used to estimate GFR based on serum creatinine, weight, and gender. eGFRcg = (140 - age in years) x (body weight in kg) x (0.85 if female) divided by 72 x serum creatinine in mg/dL.
  Moderate renal impairment= 30 mL/min ≤ eGFRCG ≤ 59 mL/min Severe renal impairment= 15 mL/min ≤ eGFRCG < 30 mL/min Change from baseline was calculated as the value at Week 24 minus the value at Baseline.
Time Frame: Baseline, Week 24
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part B: Hepatic Impairment
Number analyzed (Participants) | 77 | 31
mL/min | -0.4 [-3.9 to 4.5] | 1.9 [-5.6 to 12.2]

9. Secondary Outcome: Change From Baseline in eGFRcg in Participants With Moderate or Severe Renal Impairment and Hepatically Impaired Participants at Week 48
Description: GFR is a measure of the rate at which blood is filtered by the kidney. Cockcroft-Gault is an equation (calculation) used to estimate GFR based on serum creatinine, weight, and gender. eGFRcg = (140 - age in years) x (body weight in kg) x (0.85 if female) divided by 72 x serum creatinine in mg/dL.
  Moderate renal impairment= 30 mL/min ≤ eGFRCG ≤ 59 mL/min Severe renal impairment= 15 mL/min ≤ eGFRCG < 30 mL/min Change from baseline was calculated as the value at Week 48 minus the value at Baseline.
Time Frame: Baseline, Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part B: Hepatic Impairment
Number analyzed (Participants) | 73 | 31
mL/min | -0.5 [-4.1 to 3.0] | 1.2 [-13.5 to 6.5]

10. Secondary Outcome: Change From Baseline in eGFRcg in Participants With Moderate or Severe Renal Impairment and Hepatically Impaired Participants at Week 96
Description: GFR is a measure of the rate at which blood is filtered by the kidney. Cockcroft-Gault is an equation (calculation) used to estimate GFR based on serum creatinine, weight, and gender. eGFRcg = (140 - age in years) x (body weight in kg) x (0.85 if female) divided by 72 x serum creatinine in mg/dL.
  Moderate renal impairment= 30 mL/min ≤ eGFRCG ≤ 59 mL/min Severe renal impairment= 15 mL/min ≤ eGFRCG < 30 mL/min Change from baseline was calculated as the value at Week 96 minus the value at Baseline.
Time Frame: Baseline, Week 96
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part B: Hepatic Impairment
Number analyzed (Participants) | 66 | 25
mL/min | 1.0 [-2.8 to 4.5] | -2.4 [-11.4 to 10.7]

11. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 24
Description: Percent change = Change from baseline at a postbaseline visit/baseline * 100%.
Time Frame: Baseline, Week 24
Population: Participants in the Hip Dual-Energy X-Ray Absorptiometry (DXA) Analysis Set (all participants who were enrolled and received at least 1 dose of study drug and had non-missing baseline hip BMD values) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 74 | 15 | 31
percent change | 0.135 (1.8348) | 0.322 (2.1835) | 0.322 (2.5105)

12. Secondary Outcome: Percent Change From Baseline in Hip BMD at Week 48
Description: Percent change = Change from baseline at a postbaseline visit/baseline * 100%.
Time Frame: Baseline, Week 48
Population: Participants in Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 72 | 14 | 31
percent change | 0.565 (2.6160) | -1.075 (3.6355) | -0.221 (3.0158)

13. Secondary Outcome: Percent Change From Baseline in Hip BMD at Week 96
Description: Percent change = Change from baseline at a postbaseline visit/baseline * 100%.
Time Frame: Baseline, Week 96
Population: Participants in Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 59 | 13 | 24
percent change | 0.425 (2.8381) | -0.834 (4.7171) | 0.277 (3.2549)

14. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 24
Description: Percent change = Change from baseline at a postbaseline visit/baseline * 100%.
Time Frame: Baseline, Week 24
Population: Participants in the Spine DXA Analysis Set (all participants who were enrolled and received at least 1 dose of study drug and had non-missing baseline spine BMD values) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 76 | 15 | 31
percent change | 1.229 (3.4252) | 0.683 (3.1370) | 1.258 (2.3416)

15. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48
Description: Percent change = Change from baseline at a postbaseline visit/baseline * 100%.
Time Frame: Baseline, Week 48
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 73 | 14 | 31
percent change | 1.516 (3.7486) | 0.016 (4.1636) | 0.535 (3.4386)

16. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 96
Description: Percent change = Change from baseline at a postbaseline visit/baseline * 100%.
Time Frame: Baseline, Week 96
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 61 | 13 | 23
percent change | 1.293 (4.4136) | -0.283 (4.5327) | -0.249 (3.9127)

17. Secondary Outcome: Percentage of Participants Achieving Virologic Response (Plasma HBV DNA < 20 IU/mL) at Week 48
Description: The percentage of participants with HBV DNA < 20 IU/mL at Week 48 was determined by the Missing = Failure (M = F) approach.
Time Frame: Weeks 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants | 92.3 | 93.3 | 100.0

18. Secondary Outcome: Percentage of Participants Achieving Virologic Response (Plasma HBV DNA < 20 IU/mL) at Week 96
Description: as for outcome 17
Time Frame: Weeks 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants | 83.3 | 86.7 | 77.4

19. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 20 IU/mL and Target Detected (≥ Lower Limit of Detection [LLOD]) at Week 24
Description: The percentage of participants with HBV DNA < 20 IU/mL and target detected (≥ LLOD; i.e. 10 IU/mL) at Week 24 was determined by the M = F approach.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants | 21.8 | 40.0 | 22.6

20. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 20 IU/mL and Target Detected (≥ LLOD) at Week 48
Description: The percentage of participants with HBV DNA < 20 IU/mL and target detected (≥ LLOD; i.e. 10 IU/mL) at Week 48 was determined by the M = F approach.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants | 26.9 | 26.7 | 25.8

21. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 20 IU/mL and Target Detected (≥ LLOD) at Week 96
Description: The percentage of participants with HBV DNA < 20 IU/mL and target detected (≥ LLOD; i.e. 10 IU/mL) at Week 96 was determined by the M = F approach.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants | 14.1 | 20.0 | 0

22. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 20 IU/mL and Target Not Detected (< LLOD) at Week 24
Description: The percentage of participants with HBV DNA < 20 IU/mL and target not detected (< LLOD; i.e. 10 IU/mL) at Week 24 was determined by the M = F approach.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants | 75.6 | 60.0 | 77.4

23. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 20 IU/mL and Target Not Detected (< LLOD) at Week 48
Description: The percentage of participants with HBV DNA < 20 IU/mL and target not detected (< LLOD; i.e. 10 IU/mL) at Week 48 was determined by the M = F approach.
Time Frame: Weeks 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants | 65.4 | 66.7 | 74.2

24. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 20 IU/mL and Target Not Detected (< LLOD) at Week 96
Description: The percentage of participants with HBV DNA < 20 IU/mL and target not detected (< LLOD; i.e. 10 IU/mL) at Week 96 was determined by the M = F approach.
Time Frame: Weeks 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants | 69.2 | 66.7 | 77.4

25. Secondary Outcome: Percentage of Participants With Serological Response: Loss of Hepatitis B s-Antigen (HBsAg) at Week 24
Description: HBsAg loss was defined as HBsAg changing from positive at baseline to negative at a postbaseline. The M = F approach was used for this analysis.
Time Frame: Week 24
Population: The Serologically Evaluable Full Analysis Set for HBsAg Loss/Seroconversion (all participants who were enrolled and received at least 1 dose of study drug, and with HBsAg positive and HBsAb negative or missing at baseline) with available data were analyzed..
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 30
percentage of participants | 0 | 0 | 0

26. Secondary Outcome: Percentage of Participants With Serological Response: Loss of HBsAg at Week 48
Description: as for outcome 25
Time Frame: Week 48
Population: Participants in the Serologically Evaluable Full Analysis Set for HBsAg Loss/Seroconversion with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 30
percentage of participants | 0.0 | 6.7 | 3.3

27. Secondary Outcome: Percentage of Participants With Serological Response: Loss of HBsAg at Week 96
Description: as for outcome 25
Time Frame: Week 96
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 30
percentage of participants | 0 | 0 | 6.7

28. Secondary Outcome: Percentage of Participants With Serological Response: Seroconversion to Anti-HBs at Week 24
Description: HBsAg seroconversion was defined as HBsAg loss and HBsAb test changing from negative/missing at baseline to positive at a postbaseline visit. The M = F approach was used for this analysis.
Time Frame: Week 24
Population: The Serologically Evaluable Full Analysis Set for HBsAg Loss/Seroconversion were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 30
percentage of participants | 0 | 0 | 0

29. Secondary Outcome: Percentage of Participants With Serological Response: Seroconversion to Anti-HBs at Week 48
Description: as for outcome 28
Time Frame: Week 48
Population: Participants in the Serologically Evaluable Full Analysis Set for HBsAg Loss/Seroconversion were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 30
percentage of participants | 0 | 0 | 0

30. Secondary Outcome: Percentage of Participants With Serological Response: Seroconversion to Anti-HBs at Week 96
Description: as for outcome 28
Time Frame: Week 96
Population: The Serologically Evaluable Full Analysis Set for HBsAg Loss/Seroconversion were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 30
percentage of participants | 0 | 0 | 0

31. Secondary Outcome: Percentage of Participants With Serological Response: Loss of HBeAg in HBeAg-Positive Participants at Week 24
Description: HBeAg loss was defined as HBeAg changing from positive at baseline to negative at a postbaseline. The M = F approach was used for this analysis.
Time Frame: Week 24
Population: The Serologically Evaluable Full Analysis Set for HBeAg Loss/Seroconversion included all participants who were enrolled and received at least 1 dose of study drug, and with HBeAg positive and HBeAb negative or missing at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 13 | 3 | 3
percentage of participants | 0 | 0 | 0

32. Secondary Outcome: Percentage of Participants With Serological Response: Loss of HBeAg in HBeAg-Positive Participants at Week 48
Description: as for outcome 31
Time Frame: Week 48
Population: Participants in the Serologically Evaluable Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 13 | 3 | 3
percentage of participants | 0 | 0 | 0

33. Secondary Outcome: Percentage of Participants With Serological Response: Loss of HBeAg in HBeAg-Positive Participants at Week 96
Description: as for outcome 31
Time Frame: Week 96
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 13 | 3 | 3
percentage of participants | 0 | 33.3 | 0

34. Secondary Outcome: Percentage of Participants With Serological Response: Seroconversion to Anti-HBe in HBeAg-Positive Participants at Week 24
Description: HBeAg seroconversion was defined as HBeAg loss and HBeAb test changing from negative/missing at baseline to positive at a postbaseline visit. The M = F approach was used for this analysis.
Time Frame: Week 24
Population: The Serologically Evaluable Full Analysis Set for HBeAg Loss/Seroconversion were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 13 | 3 | 3
percentage of participants | 0 | 0 | 0

35. Secondary Outcome: Percentage of Participants With Serological Response: Seroconversion to Anti-HBe in HBeAg-Positive Participants at Week 48
Description: as for outcome 34
Time Frame: Week 48
Population: The Serologically Evaluable Full Analysis Set for HBeAg Loss/Seroconversion were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 13 | 3 | 3
percentage of participants | 0 | 0 | 0

36. Secondary Outcome: Percentage of Participants With Serological Response: Seroconversion to Anti-HBe in HBeAg-Positive Participants at Week 96
Description: as for outcome 34
Time Frame: Week 96
Population: The Serologically Evaluable Full Analysis Set for HBeAg Loss/Seroconversion were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 13 | 3 | 3
percentage of participants | 0 | 33.3 | 0

37. Secondary Outcome: Percentage of Participants With Normal Alanine Aminotransferase (ALT) at Week 24 by Central Laboratory and the American Association for the Study of Liver Diseases (AASLD) Criteria
Description: Central laboratory ULN for ALT were as follows: ≤ 43 U/L for males aged 18 to < 69 years and ≤ 35 U/L for males aged ≥ 69 years; ≤ 34 U/L for females aged 18 to < 69 years and ≤ 32 U/L for females aged ≥ 69 years. The ULN for ALT using the 2018 AASLD normal range was 25 U/L for females and 35 U/L for males. The M = F approach was used for this analysis.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants
  ALT by central laboratory | 92.3 | 93.3 | 83.9
  ALT by AASLD criteria | 87.2 | 93.3 | 80.6

38. Secondary Outcome: Percentage of Participants With Normal ALT at Week 48 by Central Laboratory and the AASLD Criteria
Description: as for outcome 37
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants
  ALT by central laboratory | 89.7 | 86.7 | 90.3
  ALT by AASLD criteria | 87.2 | 80.0 | 80.6

39. Secondary Outcome: Percentage of Participants With Normal ALT at Week 96 by Central Laboratory and the AASLD Criteria
Description: as for outcome 37
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 78 | 15 | 31
percentage of participants
  ALT by central laboratory | 82.1 | 86.7 | 71.0
  ALT by AASLD criteria | 74.4 | 86.7 | 58.1

40. Secondary Outcome: Percentage of Participants With Normalized ALT at Week 24 by Central Laboratory and the AASLD Criteria
Description: ALT normalization was defined as an ALT value that changed from above the normal range at baseline to within the normal range at the given postbaseline visit. Central laboratory ULN for ALT were as follows: ≤ 43 U/L for males aged 18 to < 69 years and ≤ 35 U/L for males aged ≥ 69 years; ≤ 34 U/L for females aged 18 to < 69 years and ≤ 32 U/L for females aged ≥ 69 years. The ULN for ALT using the 2018 AASLD normal range was 25 U/L for females and 35 U/L for males. The M = F approach was used for this analysis.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with Baseline ALT > ULN were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 5 | 0 | 10
percentage of participants
  Normalized ALT by Central Laboratory: number analyzed (Participants) | 3 | 0 | 4
  Normalized ALT by Central Laboratory | 66.7 |  | 50.0
  Normalized ALT by AASLD Criteria | 40.0 |  | 60.0

41. Secondary Outcome: Percentage of Participants With Normalized ALT at Week 48 by Central Laboratory and the AASLD Criteria
Description: as for outcome 40
Time Frame: Week 48
Population: Participants in the Full Analysis Set with Baseline ALT > ULN were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 5 | 0 | 10
percentage of participants
  Normalized ALT by Central Laboratory: number analyzed (Participants) | 3 | 0 | 4
  Normalized ALT by Central Laboratory | 33.3 |  | 75.0
  Normalized ALT by AASLD Criteria | 60.0 |  | 60.0

42. Secondary Outcome: Percentage of Participants With Normalized ALT at Week 96 by Central Laboratory and the AASLD Criteria
Description: as for outcome 40
Time Frame: Week 96
Population: Participants in the Full Analysis Set with Baseline ALT > ULN were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 5 | 0 | 10
percentage of participants
  Normalized ALT by Central Laboratory: number analyzed (Participants) | 3 | 0 | 4
  Normalized ALT by Central Laboratory | 33.3 |  | 50.0
  Normalized ALT by AASLD Criteria | 20.0 |  | 50.0

43. Secondary Outcome: Change From Baseline in FibroTest® Score at Week 24
Description: The FibroTest® score is used to assess liver fibrosis. Scores range from 0.00 to 1.00, with higher scores indicating a greater degree of fibrosis. Change from baseline was calculated as the value at Week 24 minus the value at Baseline.
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 74 | 15 | 31
units on a scale | -0.01 (0.099) | -0.01 (0.064) | -0.05 (0.106)

44. Secondary Outcome: Change From Baseline in FibroTest® Score at Week 48
Description: The FibroTest® score is used to assess liver fibrosis. Scores range from 0.00 to 1.00, with higher scores indicating a greater degree of fibrosis. Change from baseline was calculated as the value at Week 48 minus the value at Baseline.
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 73 | 14 | 31
units on a scale | -0.03 (0.102) | -0.01 (0.071) | -0.03 (0.102)

45. Secondary Outcome: Change From Baseline in FibroTest® Score at Week 96
Description: The FibroTest® score is used to assess liver fibrosis. Scores range from 0.00 to 1.00, with higher scores indicating a greater degree of fibrosis. Change from baseline was calculated as the value at Week 96 minus the value at Baseline.
Time Frame: Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease | Part B: Hepatic Impairment
Number analyzed (Participants) | 65 | 13 | 26
units on a scale | -0.01 (0.114) | 0.03 (0.107) | -0.02 (0.118)

46. Secondary Outcome: Change From Baseline in Child-Pugh-Turcotte (CPT) Score in Hepatically Impaired Participants at Week 24
Description: CPT scores grade the severity of cirrhosis and are used to determine the need for liver transplantation. Scores can range from 5 to 15, with higher scores indicating a greater severity of disease.
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set only from Part B (Hepatic Impairment) were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: Hepatic Impairment
Number analyzed (Participants) | 31
units on a scale | 0 (1.1)

47. Secondary Outcome: Change From Baseline in CPT Score in Hepatically Impaired Participants at Week 48
Description: as for outcome 46
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set only from Part B (Hepatic Impairment) were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: Hepatic Impairment
Number analyzed (Participants) | 31
units on a scale | 0 (1.1)

48. Secondary Outcome: Change From Baseline in CPT Score in Hepatically Impaired Participants at Week 96
Description: as for outcome 46
Time Frame: Baseline, Week 96
Population: Participants in the Full Analysis Set only from Part B (Hepatic Impairment) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: Hepatic Impairment
Number analyzed (Participants) | 25
units on a scale | 0 (1.2)

49. Secondary Outcome: Change From Baseline in Model for End-Stage Liver Disease (MELD) Score in Hepatically Impaired Participants at Week 24
Description: MELD scores are used to assess prognosis and suitability for liver transplantation. Scores can range from 6 to 40, with higher scores indicating greater disease severity.
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set only from Part B (Hepatic Impairment) were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: Hepatic Impairment
Number analyzed (Participants) | 31
units on a scale | -0.6 (1.94)

50. Secondary Outcome: Change From Baseline in MELD Score in Hepatically Impaired Participants at Week 48
Description: as for outcome 49
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set only from Part B (Hepatic Impairment) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: Hepatic Impairment
Number analyzed (Participants) | 30
units on a scale | 0.1 (2.35)

51. Secondary Outcome: Change From Baseline in MELD Score in Hepatically Impaired Participants at Week 96
Description: as for outcome 49
Time Frame: Baseline, Week 96
Population: Participants in the Full Analysis Set only from Part B (Hepatic Impairment) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: Hepatic Impairment
Number analyzed (Participants) | 25
units on a scale | -1.0 (1.61)

ADVERSE EVENTS:
Time Frame: Adverse Events: From the first dose date up to last dose date (maximum: 108.1 weeks) plus 3 days; All-Cause Mortality: Enrollment up to last dose date (maximum: 166.2 weeks) plus 3 days
Description: Adverse Events: The Safety Analysis Set included all participants who were enrolled and received at least 1 dose of study drug.
  All-Cause Mortality: The Full Analysis Set included all participants who were enrolled and received at least one dose of study drug.
Groups:
- Part A (Renal Impairment): End Stage Renal Disease (Cohort 2): Participants with CHB and end stage renal disease who were virologically suppressed and taking TDF), a TDF-containing anti-HBV regimen, or OAVs, switched to TAF and received TAF 25 mg tablet once daily orally for 96 weeks.
- Part B (Hepatic Impairment): Moderate or Severe Hepatic Impair: Participants with CHB and moderate or severe hepatic impairment who were virologically suppressed and taking TDF), a TDF-containing anti-HBV regimen, or OAVs, switched to TAF and received TAF 25 mg tablet once daily orally for 96 weeks.
Arm/Group | Part A (Renal Impairment): Moderate or Severe Renal Impairment | Part A (Renal Impairment): End Stage Renal Disease (Cohort 2) | Part B (Hepatic Impairment): Moderate or Severe Hepatic Impair
All-Cause Mortality (participants affected / at risk) | 2/78 | 1/15 | 2/31
Serious Adverse Events (participants affected / at risk) | 12/78 | 8/15 | 10/31
Other Adverse Events (participants affected / at risk) | 34/78 | 15/15 | 23/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (Renal Impairment): Moderate or Severe Renal Impairment (N=78) | Part A (Renal Impairment): End Stage Renal Disease (Cohort 2) (N=15) | Part B (Hepatic Impairment): Moderate or Severe Hepatic Impair (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0
Adrenal mass (Endocrine disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Catheter site discharge (General disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Fungal cystitis (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Drain site complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Carcinoembryonic antigen increased (Investigations) | 1 | 0 | 0
Model for end stage liver disease score increased (Investigations) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Focal myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 2
Ischaemic stroke (Nervous system disorders) | 2 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (Renal Impairment): Moderate or Severe Renal Impairment (N=78) | Part A (Renal Impairment): End Stage Renal Disease (Cohort 2) (N=15) | Part B (Hepatic Impairment): Moderate or Severe Hepatic Impair (N=31)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Cataract (Eye disorders) | 1 | 1 | 1
Cataract nuclear (Eye disorders) | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 1
Iridocyclitis (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 4
Constipation (Gastrointestinal disorders) | 2 | 4 | 3
Dental caries (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 6
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 3 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Chest discomfort (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 2
Oedema peripheral (General disorders) | 1 | 1 | 2
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 5
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 2
Endophthalmitis (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 6 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 3 | 6
Urinary tract infection (Infections and infestations) | 3 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 2
Bone density decreased (Investigations) | 1 | 0 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Bone loss (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Ovarian cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 2
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 1 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 3 | 1 | 1
Renal mass (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 4 | 1
Hypotension (Vascular disorders) | 0 | 2 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
Venous occlusion (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT03180619/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03180619/SAP_002.pdf